CLINICAL TRIAL: NCT01395056
Title: Study of Chemotherapy Combined With Adoptive Cellular Therapy With Dendritic and Cytokine-induced Killer Cells in Triple Negative Breast Cancer Patients
Brief Title: Study of Chemotherapy With Adoptive Cellular Therapy With DC-CIK Cells in Triple Negative Breast Cancer Patients
Acronym: DCCIK
Status: Completed | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Ren, Director of the Medical Oncology, Peking University Cancer Hospital & Institute
Other Study IDs: CTX+TSPA+CBP
Record Dates: First submitted 2011-07-14; First posted 2011-07-15 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
Keywords: breast neoplasm; Neoplasm Metastasis; Drug Therapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — about 4ml peripheral vein blood，paraffin section on metastatic tissue，
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To access the effectiveness of cyclophosphamide combined thiotepa and carboplatin chemotherapy combined with adoptive cellular therapy with dendritic and cytokine-induced killer cells in triple negative metastatic breast cancer patients

DETAILED DESCRIPTION:
1. Metastatic breast cancer patients should be definitively diagnosis based on histopathology, with ER-negative and PR-negative, FISH testing for her-2-negative
2. All the patients enrolled will be given standard cyclophosphamide combined thiotepa and carboplatin chemotherapy and cellular therapy.Cellular therapy consisting of one cycle of chemotherapy followed by an apheresis and ex vivo cultures to generate DC and CIK, followed by low-dose Oral Cyclophosphamide .
3. The response is assessed using Response Evaluation Criteria in Solid Tumor Group (RECIST) guidelines.
4. Estimate time to progression, survival rates and clinical benefit response on patients.
5. Find biomarkers associated with drug response.

ELIGIBILITY:
Inclusion Criteria:

* Failure to anthracycline and/or taxol chemotherapy;
* metastatic tumor is histologically confirmed by immunohistochemical staining to be ER-negative and PR-negative. FISH testing for her-2-negative;
* Metastatic tumor can not be removed through surgery procedure;
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* Normal cardiac, hepatic, renal and bone marrow functions;
* Life expectancy ≥3 months.

Exclusion Criteria:

* Central nervous system metastases;
* Serious or uncontrolled concurrent medical illness;
* History of other malignancies;
* Having been enrolled in some other clinal trials within a month;

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female patients with metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
progression-free survival | six months to two year
  progression-free survivalis measured from the date therapy is initiated to the date of documented disease progression or death

SECONDARY OUTCOMES:
clinical benefit response and overall survival | six months to two year
  clinical benefit response include complete release(CR), partial release (PR), stable disease (SD).

CONTACTS AND LOCATIONS:
Overall Officials: Jing Yu, MD, PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China